CLINICAL TRIAL: NCT02859974
Title: Treatment of Exertion Induced Paradoxical Vocal Fold Motion Disorder (PVFMD) With a Form of Respiratory Retraining Technique
Brief Title: Treatment of Paradoxical Vocal Fold Motion Disorder (PVFMD) With a Form of Respiratory Retraining Technique
Acronym: PVFMDRespRet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Hadas Golan, CCC-SLP Hadas Golan, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33940
Record Dates: First submitted 2016-08-03; First posted 2016-08-09 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Paradoxical Vocal Fold Motion Disorder; Vocal Cord Dysfunction
Keywords: Paradoxical vocal fold motion disorder (PVFMD); vocal cord dysfunction (VCD); Respiratory retraining; Respiratory disorders
MeSH Terms: conditions — Vocal Cord Dysfunction; Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory retraining for PVFMD (Experimental): Single arm study
  Interventions: Behavioral: Respiratory retraining for PVFMD

INTERVENTIONS:
Behavioral: Respiratory retraining for PVFMD — Patients serve as their own controls. During a three week baseline, participants will complete the Dyspnea Index (DI), and have their heart rate, Resp. minute volume and ETCO2 on days 1 and 21 (or on the day treatment commences). Participants will complete a "daily log" reporting their daily symptoms. This will serve as the baseline "pre"phase.
  Post 1 phase will include five individual therapy sessions teaching the respiratory retraining techniques over an estimated three week period.
  Post2 phase will comprise of a six week home practice phase. There will be four measuring points per participant: pre1/pre2 measurements on day 1 and 21 (or on the day therapy begins), post1 upon completing five therapy sessions and post 2 upon completion of the home practice phase.

SUMMARY:
Paradoxical Vocal Fold Motion Disorder (PVFMD), otherwise known as vocal cord dysfunction (VCD) is a laryngeal breathing disorder that has several potential causes. In some individuals, exertion is the predominant trigger. PVFMD can present like an asthma attack, but asthma medication is ineffective in treating it. The effects of untreated PVFMD can be devastating, leading to harmful, invasive, and ineffective treatments over a period of years. Numerous anecdotal reports indicate that several behavioral techniques, may be surprisingly effective and even curative. However, data are lacking. The form of respiratory retraining technique tested in the current study educates people with PVFMD about breathing and teaches them a number of breathing exercises specially designed to restore normal breathing patterns.

This case series study will use a dyspnea perception questionnaire, patient daily logs, and physiological measurements of heart rate and breathing to examine whether this form of therapy can improve exertion-induced PVFMD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy according to available medical history or by patient and parent report on the health questionnaire
* Patients with no history of asthma, or well-controlled asthma
* A diagnosis of PVFMD by an otolaryngologist based on set criteria in-line with the National Jewish PVFMD diagnostics protocol (based on Hicks, 2008; Hoyte, 2013, Martin, 1987), to be confirmed by an additional otolaryngologist blinded to the initial diagnosis
* A score of three or more on the dyspnea index (DI)

Exclusion Criteria:

* A score of less than three on the DI
* People diagnosed with hypertension, cardiac disorders or severe pulmonary diseases which affect blood oxygen saturation
* Uncontrolled asthma

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Change in Dyspnea Index (DI) score pre and post therapy | measured at four points: day 1, day 21, day 42 and day 84
  a 10-item symptom-based questionnaire validated on individuals with upper airway pathology, including PVFMD (Gartner-Schmidt, Shembel, Zullo, & Rosen, 2014)
Change in the frequency and control of PVFMD patient-reported symptoms, pre and post therapy, measured by a daily log | Measured daily for 84 days
  The log will reflect participants' perceptions of frequency of PVFMD symptoms and their severity and ability to control them, using a three-item questionnaire using visual analogue scales (VAS) created by the investigators

SECONDARY OUTCOMES:
Change in respiratory minute volume using Spirometry pre and post therapy | Measured on day 1, 21, 42 and 84
  This measure was chosen to quantify the volume (frequency and depth) of exchanged air to determine to what extent individuals who undergo the tested respiratory retraining technique change the rate and depth of respiration.
ETCO2 using Capnometry | Measured on day 1, 21, 42 and 84
  ETCO2, or blood gas end tidal carbon dioxide, is considered a surrogate measure for arterial CO2 levels (Bowler, 1998; Gardner 1996). Increased levels of ETCO2 have been suggested to improve symptoms of hyperventilation caused by over-breathing (Courtney, 2008; Stark & Stark, 2002).
Heart rate using pulse oximetry and during home practice measured by the participants taking their pulse | Measured on day 1, 21, and then measured three times daily till day 84
  A reduction in heart rate from pre-therapy to post-therapy may suggest decreased levels of arousal, which may also correlate with respiratory minute volume.
Control Pause (CP) or Steps | measured on day 1 and 21 and then measured three times daily till day 84
  The CP/steps is a rough measure to determine the internal validity of the respiratory retraining program in the cohort with PVFMD. CP/Steps measures are proposed to be correlated with ETCO2 measurements (Stark & Stark, 2002, p.77; p. 113).

CONTACTS AND LOCATIONS:
Overall Officials: Dana Halevi-Katz, BA-SLP, Principal Investigator — University of Haifa
Locations (1):
- BUMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoyte FC. Vocal cord dysfunction. Immunol Allergy Clin North Am. 2013 Feb;33(1):1-22. doi: 10.1016/j.iac.2012.10.010. Epub 2012 Dec 21. PMID 23337061
- [Background] Patel RR, Venediktov R, Schooling T, Wang B. Evidence-Based Systematic Review: Effects of Speech-Language Pathology Treatment for Individuals With Paradoxical Vocal Fold Motion. Am J Speech Lang Pathol. 2015 Aug;24(3):566-84. doi: 10.1044/2015_AJSLP-14-0120. PMID 25836980
- [Result] Mathers-Schmidt BA, Brilla LR. Inspiratory muscle training in exercise-induced paradoxical vocal fold motion. J Voice. 2005 Dec;19(4):635-44. doi: 10.1016/j.jvoice.2005.03.005. Epub 2005 Aug 19. PMID 16112543
- See also: Informaiton on vocal cord dysfunction by Jewish National Health — https://www.nationaljewish.org/healthinfo/conditions/Vocal-Cord-Dysfunction